CLINICAL TRIAL: NCT05538923
Title: Dental Caries, Dental Erosion and Periodontal Disease in Children With Inflammatory Bowel Disease
Brief Title: Oral Health in Children With Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Collaborators: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Other Study IDs: HDireskeneli
Record Dates: First submitted 2022-09-11; First posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Oral Health in Children With Inflammatory Bowel Disease
Keywords: inflammatory bowel disease, children, permanent dentition, nutritional habits
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with IBD: Patients with inflammatory bowel disease on remission period
  Interventions: Other: No intervention was given to the patients
- Control: Age- and gender- matched healthy population
  Interventions: Other: No intervention was given to the patients

INTERVENTIONS:
Other: No intervention was given to the patients — This study was an observational epidemiological study.

SUMMARY:
In adults with inflammatory bowel disease (IBD), a higher prevalence of dental caries and periodontal disease has been reported compared with healthy control subjects, but similar data on children are missing in the literature.We aimed to evaluate the prevalence of dental erosion, dental caries and periodontal disease in children with IBD.

DETAILED DESCRIPTION:
In this age- and gender-matched prospective case-control study, detailed questionnaires including nutritional habits and oral examinations were completed for 32 IBD patients aged 11 to 18 (15,53±2,00 yr) and 32 healthy controls based on the established criteria of the World Health Organization by the same pediatric dentist.

ELIGIBILITY:
Inclusion Criteria:

* 11-18 years of age
* Study population with IBD in the remission period of disease
* Permanent dentition stage

Exclusion Criteria:

* Those who refused or whose families refused participation in this study
* Study population with IBD in the active period of disease
* Primary or mix dentition stage
* Systemic conditions, or medications with impact on periodontal tissues and previous orthodontic or periodontal treatment within the last year.
* Smoking

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Study population with inflammatory bowel disease in the remission period.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Dental caries | In one year
  In the present study WHO criteria were used to detect DMFT (decayed, missing and filled permanent teeth) scores
Dental erosion | In one year
  Dental erosion status was determined with the basic erosive wear examination (BEWE) index
Periodontal disease | In one year
  The patients' and controls' gingival condition was also scored according to the criteria of a Gingival Index (GI) System. The oral hygiene status was determined with the PCR index in order to assess the presence or absence of marginal plaque. The prevalence and the severity of periodontal disease were recorded with the CPITN after dividing the oral cavity into sextants.
Oral extraintestinal manifestations (EIMs) | In one year
  including the lip mucosa, buccal mucosa, gingiva; the palatal mucosa and oropharynx; the tongue dorsum, tongue ventrum, and floor of the mouth

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)